CLINICAL TRIAL: NCT02995304
Title: Preemptive Analgesia for Post Tonsillectomy Pain With IV Morphine in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Soliman Fakeeh Hospital (Other)
Responsible Party: Principal Investigator, Dr. Amr Aly Ismail Keera, Principle investigator, Dr. Soliman Fakeeh Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 03/IRB/2016
Record Dates: First submitted 2016-11-02; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Preoperative Sedation; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine and Midazolam premedication (Active Comparator): 30 children will receive 0.025 mg/kg midazolam IV followed by 0.1 mg/kg morphine 20 to 30 min before surgical incision.
  Interventions: Drug: Morphine premedication; Drug: Midazolam premedication
- Midazolam only premedication (Active Comparator): 30 children who will receive 0.025 mg/kg midazolam IV followed by saline 20 to 30 min before surgical incision.
  Interventions: Drug: Midazolam premedication; Drug: Saline premedication (placebo)

INTERVENTIONS:
Drug: Morphine premedication — 30 children will 0.1 mg/kg morphine as a premedication 20 to 30 min before surgical incision.
  Arms: Morphine and Midazolam premedication
Drug: Midazolam premedication — All children who will receive 0.025 mg/kg midazolam IV as a premedication 20 to 30 min before surgical incision.
Drug: Saline premedication (placebo) — 30 children in midazolam only group will receive saline after midazolam
  Arms: Midazolam only premedication

SUMMARY:
In this double blind study, after taking an informed consent, 60 children aged between 7 and 12 years old assigned for tonsillectomy with or without adenoidectomy will be randomly divided into three groups. The first group 30 children will receive 0.025 mg/kg midazolam IV followed by 0.1 mg/kg morphine as a premedication 20 to 30 min before surgical incision. In the second group30 children who will receive the same dose of midazolam followed by saline premedication. All groups will be compared for pain score using visual analog scale (VAS) after recovery and hourly for 8 hours and during first drinking. Heart rate (HR), blood pressure and peripheral oxygen saturation (SPO2) will be recorded before premedication, every 10 min after premedication then every 5 min during and after anesthesia. 6 point sedation score and 4 points behavioral score will be monitored every 5 min after sedation. Four-point wake-up score will be recorded every 5 min. Time of first analgesic requirement and total morphine consumption during the first post-operative 8 hours will be recorded.

DETAILED DESCRIPTION:
Tonsillectomy is a minor procedure but it causes sever post-operative pain. This pain is difficult to be controlled with opioids because the fear from respiratory depression in pediatric age group with postoperative oral bleeding. The World Heath Organization (WHO) guidelines clearly state that fear and lack of knowledge regarding the use of opioids in children should not be a barrier for effective analgesia (1). ). However, these procedures are usually day case and the use of oral morphine at home may be risky in some groups of this population (2). So decrease the analgesic requirements following these procedures will increase both satisfaction and safety. The trials for the use of morphine as a preemptive analgesia, in awake patient, have been limited to intramuscular (IM) or oral use which has a slow onset and unpredictable absorption. The use of preoperative IV morphine is not popular because of the unpleasant sensations following its administration. I will use small dose midazolam 0.025 gm/kg before morphine to prevent this sensation. In this double blind study, after taking an informed consent, 60 children aged between 7 and 12 years old assigned for tonsillectomy with or without adenoidectomy will be randomly divided into three groups. The first group 30 children will receive 0.025 mg/kg midazolam IV followed by 0.1 mg/kg morphine as a premedication 20 to 30 min before surgical incision. In the second group30 children who will receive the same dose of midazolam followed by saline premedication. Inhalational anesthesia with sevoflurane and nitrous oxide will be used in all patients. Exclusion criteria are those with bronchial asthma, obstructive sleep apnea, allergy to medications used in the study and those who are unfit for surgery or anesthesia for any reason like coagulopathy or chest infection.

All groups will be compared for pain score using visual analog scale (VAS) after recovery and hourly for 8 hours and during first drinking. HR, blood pressure and SPO2 will be recorded before premedication, every 10 min after premedication then every 5 min during and after anesthesia. 6 point sedation score and 4 points behavioral score will be monitored every 5 min after sedation. Four-point wake-up score will be recorded every 5 min. Time of first analgesic requirement and total morphine consumption during the first post-operative 8 hours will be recorded. Base line oxygen saturation, incidence of postoperative hypoxia, bleeding, nausea and vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy procedures in
* Children aged between 7 and 12 years old.

Exclusion Criteria:

Bronchial asthma, obstructive sleep apnea, allergy to medications used in the study and those who are unfit for surgery or anesthesia for any reason like coagulopathy or chest infection.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine requirement | 8 hours

SECONDARY OUTCOMES:
Postoperative nonsteroidal analgesic requirements | two days
Preoperative behavior score | 15 to 30 minutes
  B. Behavior scores:
  1 - Calm and cooperative 2 - Anxious but can be reassured 3 - Anxious and can not be reassured 4 - Crying, or resisting C. Wake-up behavior scores 1 - Calm and cooperative 2 - Not calm but could be easily calmed 3 - Not easily calmed, moderately agitated or restless 4 - Combative, excited, disoriented.
Wake-up behavior scores | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Keera, MD, Principal Investigator — Doctor Soliman Fakeeh Hospital
Locations (1):
- Doctor Soliman Fakeeh Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No